CLINICAL TRIAL: NCT06105957
Title: Addressing Rural Health Disparities by Optimizing "High Touch" Intervention Components in Digital Obesity Treatment
Brief Title: Optimal Digital Weight Loss Treatment for Rural Individuals
Acronym: iREACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: University of Virginia (Other); University of Vermont (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Delia Smith West, Professor, University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00123003; 1R01DK135227-01 (NIH)
Record Dates: First submitted 2023-10-02; First posted 2023-10-30 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obesity
Keywords: behavioral weight control; weight management; online weight loss program
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Core+Facilitated Weekly Group Sessions+Counselor Crafted Feedback+Individual Coaching Calls (Experimental): Behavioral: Core The core intervention will include 24 online weekly behavioral modules, an online interactive discussion board, a physical activity tracker, an e-scale with recommendations for daily self-weighing, dietary self-monitoring via an app, as well as weekly calorie and physical activity goals.
  Behavioral: Facilitated Weekly Group Sessions Participants will receive 24, 60-minute facilitated online video-conference-based weekly group sessions.
  Behavioral: Counselor Crafted Feedback Participants will receive up to 24 weekly messages that are crafted by a trained professional based on their dietary, physical activity, and weight monitoring for the week as well as their completion of online modules, to construct an individualized feedback message.
  Behavioral: Individual Coaching Calls Participants will receive 3 30-minute online one-on-one coaching calls to focus on identifying and addressing challenges to successful behavior change and weight loss.
  Interventions: Behavioral: Core; Behavioral: Facilitated Weekly Group Sessions; Behavioral: Counselor Crafted Feedback; Behavioral: Individual Coaching Calls
- Core+Facilitated Weekly Group Sessions+Pre-Scripted Feedback (Experimental): Behavioral: Core The core intervention will include 24 online weekly behavioral modules, an online interactive discussion board, a physical activity tracker, an e-scale with recommendations for daily self-weighing, dietary self-monitoring via an app, as well as weekly calorie and physical activity goals.
  Behavioral: Facilitated Weekly Group Sessions Participants will receive 24, 60-minute facilitated online video-conference-based weekly group sessions.
  Behavioral: Pre-Scripted Feedback Participants will receive up to 24 weekly messages constructed from a bank of pre-scripted messages that align with success, partial success, or absence of self-monitoring related to diet monitoring, physical activity, and self-weighing, as well as on weekly module engagement.
  Interventions: Behavioral: Core; Behavioral: Facilitated Weekly Group Sessions; Behavioral: Pre-Scripted Feedback
- Core+Facilitated Weekly Group Sessions+Pre-Scripted Feedback+Individual Coaching Calls (Experimental): Behavioral: Core The core intervention will include 24 online weekly behavioral modules, an online interactive discussion board, a physical activity tracker, an e-scale with recommendations for daily self-weighing, dietary self-monitoring via an app, as well as weekly calorie and physical activity goals.
  Behavioral: Facilitated Weekly Group Sessions Participants will receive 24, 60-minute facilitated online video-conference-based weekly group sessions.
  Behavioral: Pre-Scripted Feedback Participants will receive up to 24 weekly messages constructed from a bank of pre-scripted messages that align with success, partial success, or absence of self-monitoring related to diet monitoring, physical activity, and self-weighing, as well as on weekly module engagement.
  Behavioral: Individual Coaching Calls Participants will receive 3 30-minute online one-on-one coaching calls to focus on identifying and addressing challenges to successful behavior change and weight loss.
  Interventions: Behavioral: Core; Behavioral: Facilitated Weekly Group Sessions; Behavioral: Individual Coaching Calls; Behavioral: Pre-Scripted Feedback
- Core+Facilitated Weekly Group Sessions+Counselor Crafted Feedback (Experimental): Behavioral: Core The core intervention will include 24 online weekly behavioral modules, an online interactive discussion board, a physical activity tracker, an e-scale with recommendations for daily self-weighing, dietary self-monitoring via an app, as well as weekly calorie and physical activity goals.
  Behavioral: Facilitated Weekly Group Sessions Participants will receive 24, 60-minute facilitated online video-conference-based weekly group sessions.
  Behavioral: Counselor Crafted Feedback Participants will receive up to 24 weekly messages that are crafted by a trained professional based on their dietary, physical activity, and weight monitoring for the week as well as their completion of online modules, to construct an individualized feedback message.
  Interventions: Behavioral: Core; Behavioral: Facilitated Weekly Group Sessions; Behavioral: Counselor Crafted Feedback
- Core+ Counselor Crafted Feedback+Individual Coaching Calls (Experimental): Behavioral: Core The core intervention will include 24 online weekly behavioral modules, an online interactive discussion board, a physical activity tracker, an e-scale with recommendations for daily self-weighing, dietary self-monitoring via an app, as well as weekly calorie and physical activity goals.
  Behavioral: Counselor Crafted Feedback Participants will receive up to 24 weekly messages that are crafted by a trained professional based on their dietary, physical activity, and weight monitoring for the week as well as their completion of online modules, to construct an individualized feedback message.
  Behavioral: Individual Coaching Calls Participants will receive 3 30-minute online one-on-one coaching calls to focus on identifying and addressing challenges to successful behavior change and weight loss.
  Interventions: Behavioral: Core; Behavioral: Counselor Crafted Feedback; Behavioral: Individual Coaching Calls
- Core+ Counselor Crafted Feedback (Experimental): Behavioral: Core The core intervention will include 24 online weekly behavioral modules, an online interactive discussion board, a physical activity tracker, an e-scale with recommendations for daily self-weighing, dietary self-monitoring via an app, as well as weekly calorie and physical activity goals.
  Behavioral: Counselor Crafted Feedback Participants will receive up to 24 weekly messages that are crafted by a trained professional based on their dietary, physical activity, and weight monitoring for the week as well as their completion of online modules, to construct an individualized feedback message.
  Interventions: Behavioral: Core; Behavioral: Counselor Crafted Feedback
- Core+Pre-Scripted Feedback+Individual Coaching Calls (Experimental): Behavioral: Core The core intervention will include 24 online weekly behavioral modules, an online interactive discussion board, a physical activity tracker, an e-scale with recommendations for daily self-weighing, dietary self-monitoring via an app, as well as weekly calorie and physical activity goals.
  Behavioral: Pre-Scripted Feedback Participants will receive up to 24 weekly messages constructed from a bank of pre-scripted messages that align with success, partial success, or absence of self-monitoring related to diet monitoring, physical activity, and self-weighing, as well as on weekly module engagement.
  Behavioral: Individual Coaching Calls Participants will receive 3 30-minute online one-on-one coaching calls to focus on identifying and addressing challenges to successful behavior change and weight loss.
  Interventions: Behavioral: Core; Behavioral: Individual Coaching Calls; Behavioral: Pre-Scripted Feedback
- Core+Pre-Scripted Feedback (Experimental): Behavioral: Core The core intervention will include 24 online weekly behavioral modules, an online interactive discussion board, a physical activity tracker, an e-scale with recommendations for daily self-weighing, dietary self-monitoring via an app, as well as weekly calorie and physical activity goals.
  Behavioral: Pre-Scripted Feedback Participants will receive up to 24 weekly messages constructed from a bank of pre-scripted messages that align with success, partial success, or absence of self-monitoring related to diet monitoring, physical activity, and self-weighing, as well as on weekly module engagement.
  Interventions: Behavioral: Core; Behavioral: Pre-Scripted Feedback

INTERVENTIONS:
Behavioral: Core — The core intervention will include 24 online weekly behavioral modules, an online interactive discussion board, a physical activity tracker, an e-scale with recommendations for daily self-weighing, dietary self-monitoring via an app, as well as weekly calorie and physical activity goals. Weekly tips and discussion board postings invite participants to apply skills introduced in the modules and prompt interaction and social support within the closed group which starts the program simultaneously.
Behavioral: Facilitated Weekly Group Sessions — Participants will receive 24 facilitated online video-conference-based weekly group sessions. These groups will be 60 minutes long and will be facilitated by a trained professional, who reinforces the information and behavioral strategies introduced in the weekly modules, elicits the experiences of participants in applying behavioral skills to establish new diet and exercise habits, and guides problem solving. Group cohesion to offer social support is promoted.
  Arms: Core+Facilitated Weekly Group Sessions+Counselor Crafted Feedback; Core+Facilitated Weekly Group Sessions+Counselor Crafted Feedback+Individual Coaching Calls; Core+Facilitated Weekly Group Sessions+Pre-Scripted Feedback; Core+Facilitated Weekly Group Sessions+Pre-Scripted Feedback+Individual Coaching Calls
Behavioral: Counselor Crafted Feedback — Participants will receive up to 24 weekly messages that are crafted by a trained professional based on their dietary, physical activity, and weight monitoring for the week as well as their completion of online modules, to construct an individualized feedback message. The emailed feedback will provide positive reinforcement for successful goal achievement, identify possible areas for improvement, and suggest possible strategies for identified challenges.
  Arms: Core+ Counselor Crafted Feedback; Core+ Counselor Crafted Feedback+Individual Coaching Calls; Core+Facilitated Weekly Group Sessions+Counselor Crafted Feedback; Core+Facilitated Weekly Group Sessions+Counselor Crafted Feedback+Individual Coaching Calls
Behavioral: Individual Coaching Calls — Participants will receive 3 online one-on-one coaching calls to focus on identifying and addressing challenges to successful behavior change and weight loss. The first call will emphasize amplifying motivation and promoting early treatment engagement by establishing rapport, exploring personal reasons for weight loss and lifestyle change, and reinforcing and expanding change talk, and it will occur prior to starting the core program. Subsequent calls will use a motivational interviewing-informed approach to problem solve barriers to self-monitoring, particularly dietary self-monitoring because of the strong role it plays in promoting better weight loss and will occur during the first half of the program, reflecting the critical role of early engagement in the treatment program on long term weight loss success. Coaching calls will be of approximately 30 min duration and will follow a semi-structured interview format.
  Arms: Core+ Counselor Crafted Feedback+Individual Coaching Calls; Core+Facilitated Weekly Group Sessions+Counselor Crafted Feedback+Individual Coaching Calls; Core+Facilitated Weekly Group Sessions+Pre-Scripted Feedback+Individual Coaching Calls; Core+Pre-Scripted Feedback+Individual Coaching Calls
Behavioral: Pre-Scripted Feedback — Participants will receive up to 24 weekly messages constructed from a bank of pre-scripted messages that align with success, partial success, or absence of self-monitoring within each of the following domains: dietary monitoring, physical activity monitoring, and self-weighing, as well as on weekly module completion. Feedback is automatically generated based on decision algorithms and will be sent from program staff.
  Arms: Core+Facilitated Weekly Group Sessions+Pre-Scripted Feedback; Core+Facilitated Weekly Group Sessions+Pre-Scripted Feedback+Individual Coaching Calls; Core+Pre-Scripted Feedback; Core+Pre-Scripted Feedback+Individual Coaching Calls

SUMMARY:
Over 130 million adults in the US experience overweight and obesity, and rural communities experience significantly higher rates of obesity and related chronic diseases. Although lifestyle interventions successfully produce clinically significant weight losses, the availability of weight management programs is limited in rural areas. Digital interventions offer an attractive alternative for delivering lifestyle programs to rural populations. However, in-person behavioral obesity treatment programs achieve better weight losses than digital programs, likely because in-person programs typically include personnel-intensive "high touch" treatment components. Some studies indicate that having a human "behind the curtain" of a digital program through emailed feedback or with the addition of online group sessions can significantly increase weight loss. Therefore, the aims of this study are to increase the public health impact of digital obesity treatment for rural populations by simultaneously investigating 3 "high touch" intervention components. The investigators will conduct a highly efficient experiment with participants residing in non-urban areas recruited online from across the United States. Participants (N=616; 22% racial/ethnic minority; 40% male) will be randomized to: (1) weekly facilitated synchronous group video sessions (yes vs. no); (2) type of self-monitoring feedback received (counselor-crafted vs. pre-scripted); and (3) individual coaching calls (yes vs. no). These components will be layered onto our 24-week evidence-based, interactive digital weight loss program delivered to groups of eligible individuals. Based on the results of the experiment, The investigators will identify an optimized program in which each component (or combination of components) contributes meaningfully (at least 1.5 kg greater weight loss at 6-months) to enhanced weight loss. The investigators will also exploratory analyses of weight trajectories 6-months post-treatment (i.e., at 12-months) to elucidate extended impact of the specific components on weight control. Ultimately, this research will set the stage for confirming the most promising digital behavioral weight loss intervention that can be used without geographic borders to reduce obesity rates among rural residents and provide the evidence needed to establish best practice policies for broadly effective digital approaches to weight control.

ELIGIBILITY:
Inclusion Criteria:

* have a body mass index [BMI] > 25-55 kg/m2;

  * home address in a zip code classified as non-urban; classification of an individual as living in a non-urban area will be determined by meeting any one of the following criteria: (1) having a home address corresponding to a Rural-Urban Commuting Area [RUCA] code of 4-10); (2) qualifying as rural under the Centers for Medicare and Medicaid Services Rural Health Clinic Program based on the 2010 or 2020 Census Bureau data; or (3) meeting the definition of rural from the Federal Office of Rural Health Policy;
  * have no physical limitations that prevent walking at a moderate pace for at least 10 minutes without stopping;
  * be able to provide informed consent;
  * have access to a smartphone and a computer or tablet with a video camera and stable access to the Internet (at home or work or some other stable source of access);
  * complete all screening and baseline questionnaires and activities.

Exclusion Criteria:

* only one member of a household may participate concurrently.
* currently participating in another weight loss program, taking a weight loss medication, have a history of bariatric surgery, or lost ≥ 10 pounds during the past 6-months;
* are pregnant, lactating, less than 6 months post-partum, or plan to become pregnant during the time frame of the investigation;
* report a medical condition that would affect the safety and/or efficacy of a weight management program involving diet and physical activity (e.g., uncontrolled heart condition, dementia, bulimia nervosa or binge eating disorder, or other significant psychiatric problems);
* or report conditions that in the judgment of the one of the Principal Investigators (MPIs) would render them unlikely to be able to independently follow the intervention protocol for 6 months, including conditions which might comprise their ability to engage independently with the intervention website materials, provide self-monitoring information on a smartphone app, attend Zoom video group or individual sessions at the available times (if randomized to receive these treatment components), and complete online questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in weight at 6 months | 6 months
  The difference in weight between the randomization weight and the 6 month weight. Weight values will be obtained by an electronic scale provided to participants which transmits the data to the study server.

SECONDARY OUTCOMES:
Change in weight at 12 months | 12 months
  The difference in weight between the randomization weight and the 12 month weight. Weight values will be obtained by an electronic scale provided to participants which transmits the data to the study server.

OTHER OUTCOMES:
Change in weight at 2 months | 2 months
  The difference in weight between the randomization weight and the 2 month data collection weight will be obtained by a Fitbit e-scale and transmitted to the study.server
Days of self-monitoring of body weight | Calculated continuously for 12 months
  Body Weight self-monitoring will be objectively measured as the number of days on which data on weight were transmitted via the study provided e-scale to the study team via Fitbit API
Days of dietary self-monitoring | Calculated continuously for 12 months
  Dietary self-monitoring will be objectively measured as the number of days on which data on dietary intake (foods and beverages consumed) for a minimum of 2 meals were entered into the Fitbit app and transmitted to the study team via Fitbit API
Days of physical activity self-monitoring | Calculated continuously for 12 months
  physical activity self-monitoring will be objectively measured as the number of days on which activity data were collected by wearing the study-provided Fitbit tracker and were transmitted to the study team via Fitbit API; days with wear time of a minimum of >/= 10 hours, assessed as 10 hours of non-zero heart rate measurements captured by the Fitbit device, will be considered as a day of self monitoring
Proportion of interactive, e-learning modules completed | Calculated continuously for 6 months
  The proportion of modules presenting behavioral weight management skill building lessons which are completed by participants will be determined through website utilization data and proportion completed will be calculated as number of modules completed / 24 [i.e., the total number of modules made available over the course of the intervention]
Proportion of Group Chat Sessions and Individual Coaching calls attended (percentage), for those who are randomized to receive these treatment elements | Calculated continuously for 6 months
  Attendance at treatment sessions will be recorded by interventionist personnel delivering the sessions for those participants randomized to receive these treatment elements and the proportion attended will be calculated (attended /number offered).
Self-regulation | administered at baseline, 6 and 12 months
  Self-regulation is the general ability to regulate behavior to achieve desired future outcomes and personal goals through monitoring progress through self-monitoring, goal setting, getting feedback, making adjustments to behavior, and self-rewarding; utilization of weight management self regulation processes will be assessed using the Self-Regulation Questionnaire (Kliemann, Beeken, Wardle, 2016). The measure has 63 items which are answered on a 5-point Likert scale (1-strongly disagree top 5= strong agree) and higher scores indicate a greater-self-regulation capacity.
Supportive Accountability | administered at 2 and 6 months
  Supportive accountability may increase treatment adherence when a trustworthy and caring person with specific expertise is perceived to be monitoring one's actions, and individuals feel an obligation to deliver on a commitment or explain reasons for failing to achieve an outcome. The investigators will assess supportive accountability using the Support Accountability Inventory (Meyerhoff, Haldar, & Mohr, 2021). This inventory consists of 6 items with a Likert scale response format ranging from 1 (Strongly Disagree) to 7 (Strongly Agree), with higher total scores indicating higher perceived supportive accountability
Problem solving | administered at baseline and 6 months
  Problem solving is a formal process to identify barriers and challenges to behavior change and constructively identify potential resolutions to minimize the negative impact of the barriers on behavior change; problem solving will be assessed by the Problem Solving Test (Nezu, Nezu & D'Zurilla, 2012)
Motivation | administered at baseline and 2, 6 and 12 months
  Autonomous reasons for engaging in weight control efforts (personal reasons for change or motivations that reflect an internalized rationale for change) and controlled motivation reasons for behavior change and weight loss that are externally imposed or arise from others) will be assessed with the Treatment Self-Regulation Questionnaire (Williams et al, 1996). The measure consists of 12 items, all scored using a 7-point Likert scale (1= not at all true to 7 = very true). Higher scores on the Autonomous Subscale (6 items) indicate greater autonomous motivations for behavior change and higher scores on the Controlled Motivations subscale (6 items) indicate higher controlled regulation.
Social Support for Weight Control Behaviors | administered at baseline and 2, 6 and 12 months
  Social support can facilitate weight loss and a group based program such as this can offer social support, assessed by the Social Support for Healthy Behaviors Scale which queries about social support for and sabotage of weight control behaviors from family, friends, and group members. Eighteen items assess support/sabotage for consuming a healthy dietary pattern over the previous month (the same 9 items rated separately for family members and for friends/group members using response options on a 4-point scale which ranges from almost never to almost always). Responses are coded into a social support subscale and a sabotage subscale, with higher mean scores indicating more support or more sabotage, respectively. An additional 18 items assess social support/sabotage for physical activity from family and friends using the same format (Ball & Crawford, 2006; Kiernan et al, 2012)
Group Cohesion and Social Support | administered at 2 and 6 months
  Perceived social support and group cohesion may differ based on whether individuals participate in synchronous face-to-face group sessions or if they have asynchronous, text-based communication to offer social support; therefore, we will assess group cohesion using the Group Cohesion Scale (Procidano &Heller 1983). This measure has 20 items focused on perceptions of other group members which employ a yes/no answer format plus a rating of perceived support from group leader item which ranges from 1 to 10 (with 10 being extremely supportive and 1 being not at all supportive). Higher total scores indicate greater perceived cohesion and social support from the group.
Cost | Calculated continuously for 6 months
  The non-research related costs associated with delivery of each treatment component will be continuously monitored.
Perceptions of Accountability | administered at 2 and 6 months
  Perceived accountability will be assessed using the Perceptions of Accountability subscale of the Supportive Accountability Measure (Chhabria, Ross & Leahey, 2020). This measure includes 10 items, using a 7-point Likert scale (1 = not at all to 7 i= very much). The minimum score obtainable is 10 and the highest possible score is 70, and higher scores indicate greater perceived accountability.

CONTACTS AND LOCATIONS:
Overall Officials: Delia West, PhD, Principal Investigator — University of South Carolina; Rebecca Krukowski, PhD, Principal Investigator — University of Virginia School of Medicine
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the first article reporting the primary outcomes and the first paper reporting the secondary outcomes will be shared after deidentification (text, tables, figures and appendices). Study protocol, informed consent form, statistical analysis plan and analytic code will be also available to be shared. The data will be made available 12 months after the publication of the article that reported the data. Data will be made available at the following website: https://dataverse.lib.virginia.edu/.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be made available 12 months after the publication of the article that reported the data.
Access Criteria: Data will be made available at the following website: https://dataverse.lib.virginia.edu/.
URL: http://dataverse.lib.virginia.edu

REFERENCES:
- [Background] Chhabria K, Ross KM, Sacco SJ, Leahey TM. The Assessment of Supportive Accountability in Adults Seeking Obesity Treatment: Psychometric Validation Study. J Med Internet Res. 2020 Jul 28;22(7):e17967. doi: 10.2196/17967. PMID 32720911
- [Background] Kiernan M, Moore SD, Schoffman DE, Lee K, King AC, Taylor CB, Kiernan NE, Perri MG. Social support for healthy behaviors: scale psychometrics and prediction of weight loss among women in a behavioral program. Obesity (Silver Spring). 2012 Apr;20(4):756-64. doi: 10.1038/oby.2011.293. Epub 2011 Oct 13. PMID 21996661
- [Background] Kliemann N, Beeken RJ, Wardle J, Johnson F. Development and validation of the Self-Regulation of Eating Behaviour Questionnaire for adults. Int J Behav Nutr Phys Act. 2016 Aug 2;13:87. doi: 10.1186/s12966-016-0414-6. PMID 27484457
- [Background] Mohr DC, Cuijpers P, Lehman K. Supportive accountability: a model for providing human support to enhance adherence to eHealth interventions. J Med Internet Res. 2011 Mar 10;13(1):e30. doi: 10.2196/jmir.1602. PMID 21393123
- [Background] Nezu AM, Nezu CM, Perri MG. Problem-solving therapy for depression: Theory, research and clinical guidelines. John Wiley & Sons, 1989.
- [Background] Procidano ME, Heller K. Measures of perceived social support from friends and from family: three validation studies. Am J Community Psychol. 1983 Feb;11(1):1-24. doi: 10.1007/BF00898416. PMID 6837532
- [Background] Williams GC, Grow VM, Freedman ZR, Ryan RM, Deci EL. Motivational predictors of weight loss and weight-loss maintenance. J Pers Soc Psychol. 1996 Jan;70(1):115-26. doi: 10.1037//0022-3514.70.1.115. PMID 8558405